CLINICAL TRIAL: NCT03938493
Title: Observation of the Pressure Changes of the Endotracheal Tube Cuff in the Head and Neck Surgery Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0100
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Intubation, Intratracheal
Keywords: Adults who require endotracheal intubation for head and neck surgery under general anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endotracheal intubation under general anesthesia: Adults who require endotracheal intubation for head and neck surgery under general anesthesia
  Interventions: Other: monitoring of the endotracheal tube cuff

INTERVENTIONS:
Other: monitoring of the endotracheal tube cuff — We will enroll adult patients who will undergo endotracheal intubation for general anesthesia of head and neck surgery. The cuff pressure of the endotracheal tube will be monitored continuously during anesthesia. The cuff pressure value will be recorded and analyzed after completing the study.

SUMMARY:
Endotracheal tube is a commonly used for general anesthesia in head and neck surgery. It is necessary to place the endotracheal tube in the trachea of the patient and then inflate the cuff with air. This is because the air-inflated cuff contacts the inner wall of the patient's trachea to deliver oxygen through the tube. If the cuff does not inflate, oxygen will leak through the space between the cuff and the patient's trachea. In addition, the risk of pneumonia increases. Therefore, after placing the endotracheal tube in the patient's trachea, the cuff is immediately inflated with air. However, when the cuff is inflated using an excess of air, the cuff may pressurize the mucous membrane of the tracheal wall and cause ischemia. Pressure in the over-inflated cuff was also found to be associated with post-operative sore throat, vocal cord paralysis, and nerve damage. Therefore, appropriate amount of air should be used to inflate the cuff into the air and adjust the pressure within the cuff to be within the range of 20-30 cmH2O. The authors thought that the pressure in the cuff could be changed during the operation due to various factors and that the pressure in the cuff should be monitored continuously. In this study, the investigators will monitor the cuff pressure during anesthesia and analyze the factors affecting the cuff pressure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults who require endotracheal intubation for head and neck surgery under general anesthesia

Exclusion Criteria:

* 1. Patients under 20 years old
* 2. Patients who should undergo tracheostomy
* 3. Patients who need to use an endotracheal tube without a cuff
* 4. Pregnant women
* 5. Patients who can not read the consent form or are not fluent in Korean
* 6. Patients who refused the clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who require endotracheal intubation for head and neck surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Changes of cuff pressure during anesthesia | participants will followed until post-operative 1 day.
  The investigators will monitor the pressure of the endotracheal tube cuff during anesthesia. The changes of the cuff pressure from the baseline value will be monitored continuously.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park S, Kwon YI, Kim HJ. Pressure changes in the endotracheal tube cuff in otorhinolaryngologic surgery: a prospective observational study. Front Med (Lausanne). 2023 Jun 5;10:1161566. doi: 10.3389/fmed.2023.1161566. eCollection 2023. PMID 37342495